CLINICAL TRIAL: NCT00016133
Title: A Non-Randomized Multicenter Phase I/II Study Of Active Specific Immunotherapy In Patients With Stage II and Stage III Colon Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage II or Stage III Colon Cancer That Has Been Removed During Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intracel (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: INTRACEL-ASI-2002; CDR0000068597 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-07

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — BCG Vaccine; FANG vaccine; Fluorouracil; Leucovorin; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: BCG vaccine
Biological: autologous tumor cell vaccine
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from a patient's white blood cells and tumor cells may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy combined with leucovorin and fluorouracil in treating patients who have undergone surgery to completely remove stage II or stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine safety and immunogenicity of adjuvant autologous tumor cell vaccine in patients with completely resected stage II or III adenocarcinoma of the colon.

OUTLINE: This is a multicenter study. Patients are stratified according to disease stage (II vs III).

Beginning 28-35 days after total surgical resection, patients receive adjuvant autologous tumor cell vaccine intradermally once weekly for 3 vaccinations. The first 2 vaccinations also contain BCG. Patients with stage II disease receive a fourth vaccination 6 months after surgical resection.

Beginning 10-17 days after the third vaccination, patients with stage III disease receive adjuvant leucovorin calcium IV and fluorouracil IV on days 1-5. Chemotherapy continues every 28-35 days for a total of 6 courses. These patients also receive a fourth vaccination 1 month after the completion of chemotherapy.

Patients are followed at 90 days and 6 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II or III primary adenocarcinoma of the colon

  * Completely resected within the past 28-35 days, at which time tumor tissue is harvested for vaccine production
  * No residual or metastatic disease
* No more than 1 malignant invasive primary colon cancer
* No tumor originating in the rectum (i.e., inferior tumor margin must not be at or below the peritoneal reflection)
* No perforated tumors

PATIENT CHARACTERISTICS:

Age:

* 21 to 85

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin normal
* SGOT normal
* Alkaline phosphatase normal
* No severe hepatic disease that would preclude study

Renal:

* Creatinine less than 1.5 times upper limit of normal
* No severe renal disease that would preclude study

Cardiovascular:

* No prosthetic cardiac valves
* No recent vascular prosthesis
* No postsurgical cardiovascular complication
* No severe cardiovascular disease that would preclude study

Pulmonary:

* No postsurgical pulmonary complication

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No insulin-dependent diabetes mellitus
* No severe systemic disease that would preclude study
* No congenital or acquired immune deficiency disease
* No history of chronic ulcerative colitis, Crohn's disease, Gardner's syndrome, or Turcot's syndrome
* No ileus
* No other prior malignancy except curatively treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No ongoing infection requiring systemic antibiotics
* No severe postoperative complication that would preclude study
* Carcinoembryonic antigen normal

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No other concurrent investigational immunotherapy

Chemotherapy:

* No prior systemic chemotherapy
* No other concurrent investigational chemotherapy

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* No prior radiotherapy
* No concurrent investigational radiotherapy

Surgery:

* See Disease Characteristics
* No concurrent investigational surgery

Other:

* At least 3 weeks since prior systemic antibiotic therapy of more than 5 days duration (excluding topical antibiotics or perioperative prophylactic antibiotics)
* No concurrent cytotoxic immunosuppressive agents

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Hanna Jr., PhD, Study Chair — Intracel
Locations (2):
- United States (2):
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - Inova Fairfax Hospital, Fairfax, Virginia